CLINICAL TRIAL: NCT00179153
Title: Improving The Nutritional Status Of The Malnourished Chronic Hemodialysis Patients In The State Of Tennessee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040345
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Nepro nutritional supplement

INTERVENTIONS:
Dietary Supplement: Nepro nutritional supplement — oral nutritional supplement (Nepro); every other day, 3 days per week, for 6 months

SUMMARY:
We propose to identify malnourished chronic kidney dialysis patients through a statewide effort and subsequently treat them based on a protocol (provision of oral nutritional supplementation) over a period of six (6) months.

ELIGIBILITY:
Inclusion Criteria:

* On CHD dialysis for more than 6 months
* Adequately dialyzed (Kt/V > 1.0) with a biocompatible hemodialysis membrane. Patients with Kt/V > 1.0 but < 1.4 will be evaluated for etiologies of lower than optimal dialysis dose and every effort will be made to increase the Dialysis dose to 1.4 or above. Patients with all access types will be recruited to the study.
* Suboptimal nutritional status identified by one of the following criteria:

  1. Protein catabolic rate less than 1.0 g/kg/d calculated by three-point urea kinetic modeling on at least 2 occasions over the past 3 months
  2. Progressive unintentional weight loss more than 2.5% of the initial or ideal body weight and/or patients who are less than 90% of ideal body weight.
  3. Biochemical parameters of malnutrition defined by one of the following measurements over the consecutive two months prior to inclusion:

     1. Serum albumin less than 4.0 g/dl
     2. Serum transferrin concentration less than 250 mg/dl
     3. Serum prealbumin concentration less than 32 mg/dl
  4. Subjective Global Assessment Score less than 5.

Exclusion Criteria:

* Intolerance to nutritional supplementation (unable to tolerate any of the nutritional supplements available)
* Refusal to sign a consent form
* On nutritional supplementation (IDPN or PO) within 2 weeks of the study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2005-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
increase in serum albumin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- National Kidney Foundation, Nashville, Tennessee, United States